CLINICAL TRIAL: NCT05960799
Title: Randomizes Control Trial (RCT): Superiority Study on Inter Scalene Block Execution Time for Shoulder Traumatology Surgery and Non-inferiority for Effectiveness Between Two Block Methods: Catheter Over Needle (CON) vs Catheter Through Needle (CTN).
Brief Title: Catheter Over Needle (CON) vs Catheter Through Needle (CTN).
Acronym: CONvsCTN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Alejandro Luengo, Clinical professor, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 211124003
Record Dates: First submitted 2023-06-29; First posted 2023-07-27 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Disease
Keywords: continous nerve block; peripheric nerve block; Contiplex Catheter

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Masking Description: A list of 72 names, corresponding 36 of them to contiplex C and 36 to regular contiplex will be randomized and will be introduced into sealed envelopes. Before, in order to perform the nerve block the anesthesist will open the envelope and will know wich is the catheter he has to use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contiplex C or CON (Experimental): Patients who will receive a contiplex C block for interscalene nerve block. This catheter also calls Catheter over needle (CON), wich is a catheter that is inserted at the same time that the needle is advancing.
  Interventions: Device: CON - Contiplex C™ (CC)
- Contiplex or CTN (Active Comparator): Patients who will receive a regular contiplex block for interscalene nerve block or also called Catheter throw needle (CTN). This catheter is the gold standard in this centre and the mechanism of insertion is to introduce the catheter throw the needle.
  Interventions: Device: CTN - Contiplex

INTERVENTIONS:
Device: CON - Contiplex C™ (CC) — This is a catheter used for peripherical nerve block that is inserted at the same time that the needle is being introduced. When the target is achieved, the needle is retired.
  Arms: Contiplex C or CON
Device: CTN - Contiplex — This is the traditional catheter used in this centre for peripheric nerve block. In this catheter the needle is introduced first. When the target is achieved the catheter is then introduced throw the needle and after that the needle is retired.
  Arms: Contiplex or CTN

SUMMARY:
This is a randomized clinical trial with the objective of comparing the time of insertion of two types of perineural catheters in shoulder surgery. These devices are thin lines that have to be inserted over a needle or throw a needle, depending of the type of catheter that is used. The hypothesis is: the installation of Contiplex C or catheter over needle (CON) is faster than a normal contiplex catheter or Catheter throw needle (CTN) at same rate of effectivity.

DETAILED DESCRIPTION:
In the market, there is currently two types of catheter to perform a continuous nerve block. One is called Contiplex throw needle catheter that is the most used device and other needle available for performing this block called the Contiplex® C Set, which uses a different method called Catheter over Needle (CON). This method involves advancing the catheter immediately along with the needle upon puncture, and once it reaches the target site, the needle inside the catheter is removed, leaving the catheter in its final working position. This eliminates the step of threading the catheter through the needle. Additionally, this technique allows for the visualization of the final catheter site in vivo with a single operator.

Considering the differences between both techniques, the hypothesis proposed in this study is that in adult patients undergoing shoulder and proximal humerus surgery requiring anesthetic/analgesic management with inter-scalene catheters, the use of the Catheter over Needle (CON) technique results in shorter installation time and similar effectiveness compared to the conventional technique of catheter insertion through the needle (CTN) with tunnel fixation.

The primary objectives will be to compare the block execution times between the CTN and CON techniques, as well as the effectiveness rate of both catheters

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Rotator cuff or proximal humerus surgery
* ASA I-III
* BMI 18-39 kg/m2
* Acceptance of receiving a peripheric nerve block

Exclusion Criteria:

* Inability to provide consent for the study
* Coagulopathy
* Sepsis
* Severe Renal or hepatic disease (Creatinin > 2.0 or Child C)
* Allergy to local anesthetics
* Previous peripheral nerve damage
* Refusal of postoperative continuous block technique

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-04-24 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Time of insertion | During Procedure
  The time from the insertion of the needle in the skin to: insertion of the catheter and fixation of the tegaderm in the skin

SECONDARY OUTCOMES:
Visual analogue scale (VAS). 0 (minimum) -10 (maximum) points on VAS scale. Lower scores means less pain and higher scores means more pain. | 72 hours to determinate the VAS
  compare both groups in terms of level of pain in VAS.
Rate of accidental | 72 hrs to evaluate the rate of accidental withdrawal
  Accidental withdrawal is the accidental withdrawal of the catheter before 72 hrs after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital clinico UC christus, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nogawa R, Maruyama T, Kimoto Y, Yamazaki A, Kawamata T. Comparison of catheter-over-needle and catheter-through-needle on leakage from the catheter insertion site during continuous femoral nerve block. J Anesth. 2018 Jun;32(3):439-442. doi: 10.1007/s00540-018-2479-7. Epub 2018 Mar 22. PMID 29568979
- [Background] Tsui BC, Tsui J. Less leakage and dislodgement with a catheter-over-needle versus a catheter-through-needle approach for peripheral nerve block: an ex vivo study. Can J Anaesth. 2012 Jul;59(7):655-61. doi: 10.1007/s12630-012-9713-9. Epub 2012 May 8. PMID 22565332
- [Background] Malik T, Mass D, Cohn S. Postoperative Analgesia in a Prolonged Continuous Interscalene Block Versus Single-Shot Block in Outpatient Arthroscopic Rotator Cuff Repair: A Prospective Randomized Study. Arthroscopy. 2016 Aug;32(8):1544-1550.e1. doi: 10.1016/j.arthro.2016.01.044. Epub 2016 Apr 20. PMID 27107906
- [Background] Ip VH, Rockley MC, Tsui BC. The catheter-over-needle assembly offers greater stability and less leakage compared with the traditional counterpart in continuous interscalene nerve blocks: a randomized patient-blinded study. Can J Anaesth. 2013 Dec;60(12):1272-3. doi: 10.1007/s12630-013-0032-6. Epub 2013 Sep 17. No abstract available. PMID 24043379
- [Background] Ilfeld BM. Continuous Peripheral Nerve Blocks: An Update of the Published Evidence and Comparison With Novel, Alternative Analgesic Modalities. Anesth Analg. 2017 Jan;124(1):308-335. doi: 10.1213/ANE.0000000000001581. PMID 27749354
- [Background] Tsui BC, Ip VH. Catheter-over-needle method reduces risk of perineural catheter dislocation. Br J Anaesth. 2014 Apr;112(4):759-60. doi: 10.1093/bja/aeu066. No abstract available. PMID 24645151

DOCUMENTS (1):
  • Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT05960799/Prot_000.pdf